CLINICAL TRIAL: NCT00919438
Title: Fluid Removal During Adherent Renal Monitoring
Brief Title: Non Invasive External Monitoring in Dialysis Patients
Acronym: FARM
Status: Completed | Type: Observational
Sponsor: Corventis, Inc. (Industry)
Responsible Party: Madhuri Bhat VP, Regulatory and Clinical Affairs, Corventis
Other Study IDs: COR-2008-001
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dialysis
  Interventions: Device: AVIVO™ Mobile Patient Management System

INTERVENTIONS:
Device: AVIVO™ Mobile Patient Management System — Non Invasive monitoring device
  Other Names: Diuretics- oral or IV

SUMMARY:
This is a single center, non randomized study to gather data to correlate physiological signals with the patient's fluid status during fluid removal in hemodialysis.

DETAILED DESCRIPTION:
Patients undergoing hemodialysis will be monitored with the study device . The collected information will be correlated with fluid loss.

ELIGIBILITY:
Inclusion Criteria:

* Is female or male, 18 years of age or older
* Undergoing hemodialysis for fluid removal

Exclusion Criteria:

* Is participating in another clinical study that may confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care and kidney failure clinics
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inder Anand, MD, Principal Investigator — VAMC, MN; Imad Libbus, PhD, Study Director — Corventis, Inc.